CLINICAL TRIAL: NCT02327533
Title: Gene Expression Profiles in Generalized Aggressive Periodontitis: A Gene Network-based Microarray Analysis
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Esra Guzeldemir-Akcakanat, DDS, PhD, Assoc. Prof., Kocaeli University
Other Study IDs: KOU KAEK2013/15
Record Dates: First submitted 2014-12-17; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Generalized Aggressive Periodontitis
Keywords: generalized aggressive periodontitis; microarray analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biospecimens were kept for analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Aggressive Periodontitis: The periodontal diagnosis of subjects with GAgP was established on the basis of clinical and radiographic criteria and was defined by the 1999 International World Workshop for a Classification of Periodontal Diseases and Conditions.(Lang et al., 1999)
- Controls: Control subjects had no radiographic evidence of bone loss or any sign of past and present periodontitis.

SUMMARY:
In this study, the investigators evaluated molecular biomarkers which play a role in the development of generalized aggressive periodontitis (GAgP) using gingival tissue samples through omics-based whole-genome transcriptomic while using healthy individuals as background controls.

DETAILED DESCRIPTION:
Aggressive periodontitis (AgP) is an inflammatory periodontal disease which is complex, multifactorial, and destructive. Progression and severity of the disease depend on interacting risk factors such as: immunological, microbiological, environmental, and genetic factors, as well as age, sex, and race.Some patients are genetically predisposed to AgP; they have immunological abnormalities, which are thought to be under genetic control. However, high susceptibility for periodontal destruction and the relationship between inflammatory changes, and genetic factors remain unclear.

Gene expression profiling is a powerful means of generating comprehensive genome-level data sets on diseases such as cancer, asthma, rheumatoid disorders and periodontitis, and provides significant insight information for these diseases. Gene expression profiling may provide an evidence for involving genes in the pathogenesis of AgP and generate further information other than clinical signs and symptoms of AgP.

The aim of this study was to identify gene-expression patterns of patients with generalized aggressive periodontitis by whole-transcriptome gene-expression analyses.

ELIGIBILITY:
Inclusion Criteria:

* The periodontal diagnosis of subjects with GAgP was established on the basis of clinical and radiographic criteria and was defined by the 1999 International World Workshop for a Classification of Periodontal Diseases and Conditions.(Lang et al., 1999) Patients were included if they were between 18 and 35 years of age and otherwise healthy. The bone loss estimation was radiographically performed in each patient for the assessment of the extent and severity of alveolar bone loss.

Exclusion Criteria:

* Subjects were excluded if they had any known systemic diseases or conditions that can/could influence the periodontal status (cancer, cardiovascular and respiratory diseases), any history of hepatitis and/or HIV infection, immunosuppressive chemotherapy, current pregnancy, planning a pregnancy or lactation, requirement for antibiotic prophylaxis, oral diseases other than GAgP, ongoing orthodontic therapy, a history of antibiotic therapy, or periodontal treatment within the preceding six months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Aggressive periodontitis patients: The periodontal diagnosis of subjects with GAgP was established on the basis of clinical and radiographic criteria and was defined by the 1999 International World Workshop for a Classification of Periodontal Diseases and Conditions.(Lang et al., 1999) Patients were included if they were between 18 and 35 years of age and otherwise healthy. The bone loss estimation was radiographically performed in each patient for the assessment of the extent and severity of alveolar bone loss.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
mRNA quantification | 2 months

SECONDARY OUTCOMES:
Definition of gen networking and new molecular pathways | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Esra Güzeldemir-Akçakanat, DDS, PhD, Principal Investigator — Kocaeli University

REFERENCES:
- [Background] Kinane DF, Shiba H, Hart TC. The genetic basis of periodontitis. Periodontol 2000. 2005;39:91-117. doi: 10.1111/j.1600-0757.2005.00118.x. No abstract available. PMID 16135066
- [Result] Demmer RT, Behle JH, Wolf DL, Handfield M, Kebschull M, Celenti R, Pavlidis P, Papapanou PN. Transcriptomes in healthy and diseased gingival tissues. J Periodontol. 2008 Nov;79(11):2112-24. doi: 10.1902/jop.2008.080139. PMID 18980520
- [Result] Papapanou PN, Abron A, Verbitsky M, Picolos D, Yang J, Qin J, Fine JB, Pavlidis P. Gene expression signatures in chronic and aggressive periodontitis: a pilot study. Eur J Oral Sci. 2004 Jun;112(3):216-23. doi: 10.1111/j.1600-0722.2004.00124.x. PMID 15154918